CLINICAL TRIAL: NCT06160102
Title: Appropriate Medication Use for Individuals With Intellectual Disabilities - A Matter of Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestvagoy Municipality (Other)
Collaborators: University of Oslo (Other); University of Tromso (Other)
Responsible Party: Principal Investigator, Solrun Gjertine Holm, PhD in Science of Professions, Vestvagoy Municipality
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22/658-6; Project number: 341297 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2023-10-18; First posted 2023-12-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Disabilities, Intellectual; Disability, Developmental
Keywords: Intellectual Disabilities; Developmental Disabilities; Intersectoral Collaboration; Medication Therapy Management; Medication Reconciliation; Medication Review
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Participatory action research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Framework for safe drug use in people with intellectual and/or developmental disabilities (Other): Optimizing medication management and medication therapy poses complex challenges related to the different groups, actors, and not least the data systems. To meet these challenges, we have chosen a method where the participants contribute actively in the research: participatory action research (PAR). This method involves both the action and the knowledge production being done in collaboration between all the participants, since neither the researcher nor others have exclusive right to the understanding of reality.
  Normalization process theory offers an analytical tool that helps to understand and explain the dynamic processes that occur during the implementation of complex interventions and technological and organizational innovations in health care, which includes institutional and organizational contexts and focuses on what social processes can promote and inhibit it through the integration of new routines and work forms in established social structures.
  Interventions: Other: Develop and implement the Framework for safe drug use in people with intellectual and/or developmental disabilities

INTERVENTIONS:
Other: Develop and implement the Framework for safe drug use in people with intellectual and/or developmental disabilities — Collection and analysis of drug lists and information about the users. Open / participatory observations of staff and residents during drug handling. Interviews/focus groups with residents, family, staff in the service, GPs and pharmacy staff. Interdisciplinary drug reviews based on the IMM method drug reviews, further developed by the researchers in the project.
  Design thinking. We use a design process with five stages: empathy, define, generate ideas, prototype and test. This involves user participation and experience to design the most optimal solution for the framework.
  Evaluate the framework, observations, interviews, questionnaires. Health economic evaluation.

SUMMARY:
The innovation idea is to develop valuable new knowledge about safe drug use in people with intellectual and/or developmental disabilities (IDDs). The main goal is to design a framework (routines and processes) that ensures safe drug use and provides qualitatively better services for people with IDDs. Secondary goals are that employees will experience better security when working with medicines, and interact better with people with IDD and relatives by implementing digital support functions. The innovation idea is specifically to develop/improve the following: 1) Medication management: Coordinating routines, procedures and work processes regarding all aspects of drug use, medication handling, and communication between care units for people with IDDs. 2) Medication therapy: Chart review of prescribed medication and gather knowledge about challenges related to drug use in this group. Based on this, we will develop new methods for drug reconciliation and medication reviews to optimize drug use. 3) New framework for safe drug use in the community-based services for people with IDDs.

DETAILED DESCRIPTION:
Changing, developing, and testing new routines, procedures, and communication methods for safe drug use is challenging. The complexity of systems that are involved in medication management makes it particularly challenging to create well-designed digital solutions that ensure good working procedures. The complex issues faced by people with IDDs, as well as developments within personalized medicine, means that it is crucial to build new knowledge, work in teams, and arrange for medication reconciliation and medication reviews to be carried out regularly. Furthermore, drug information must be provided, and adapted to the specific individual with an intellectual disability. In addition, the focus on personalized medicine means that the municipality must develop new guidelines for the use of pharmacogenetic tests so that the doctor can tailor drug selection and dosage to the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Users of the municipality's Service for people with disabilities

Exclusion Criteria:

-

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
To understand what is safe drug therapy and drug handling in people with intellectual and/or developmental disabilities | 12 months
  Map which drugs each patient uses and carry out medication reconciliation (nurse and pharmacist) and medication review (nurse, pharmacist and general general practitioner).
  Interviews of employees, GPs and pharmacy staff.
Formulation of multidisciplinary frameworks for optimizing drug handling and drug therapy. | 18 months
  Design thinking and co-creation of multidisciplinary frameworks
Explore usefulness of multidisciplinary frameworks | 18 months
  Transcripts of qualitative feedback. Follow-up survey of employees, GPs, pharmacy staff, and people with intellectual and/or developmental disabilities. Health economic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Wiik, MBA, Study Director — Vestvågøy Municipality
Locations (1):
- Vestvågøy Municipality, Leknes, Norway

IPD SHARING:
Plan to Share IPD: No